CLINICAL TRIAL: NCT00805688
Title: A Feasibility Study for Identifying the Role of Symptom Outcomes and Biomarkers in Survival in Patients With Metastatic Pancreatic Cancer
Brief Title: Identifying the Role of Symptom Outcomes and Biomarkers in Survival in Patients With Metastatic Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0582
Record Dates: First submitted 2008-12-05; First posted 2008-12-10 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Pancreatic Cancer
Keywords: Questionnaire; Pancreas; Pancreatic Cancer; Metastatic Disease; symptom outcomes; Biomarkers; Pedometer; MDASI-GI symptom assessment; interactive voice response telephone system; IVRS
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood drawn (around 3½ tablespoons) before treatment starts to measure cytokines (biomarkers) and DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptom Study: Questionnaires + Blood Draw + Pedometer used to learn about symptoms related to chemotherapy and the disease, in patients with advanced pancreatic cancer.
  Interventions: Behavioral: Questionnaires; Procedure: Blood Draws; Device: Pedometer

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires including symptom review (MDSAI-GI) via personal or telephone interviews (interactive voice response telephone system - IVRS)
  Other Names: survey
Procedure: Blood Draws — Blood sample (3½ tbs.)to measure levels of cytokines (biomarkers in the blood) and DNA (the genetic material in cells) before treatment starts.
Device: Pedometer — Worn daily to measure physical activity.

SUMMARY:
The goal of this clinical research study is to learn about symptoms related to chemotherapy and the disease, in patients with advanced pancreatic cancer. Researchers will study the possible reason for these symptoms by drawing blood samples and comparing the test results to the symptoms you experience. The study will also use a special telephone system for measuring the symptoms of participants during and after therapy. Your level of physical activity will also be studied using a pedometer and study diary.

DETAILED DESCRIPTION:
Researchers want to try to improve patient care for advanced pancreatic cancer by looking at how some symptoms create a great burden on daily life. They also want to find out which "markers" in the blood. Biomarkers are substances found in the blood, such as cytokines, certain proteins, and DNA changes. These biomarkers may help doctors predict "symptom burden" during therapy.

Researchers would also like to collect data about your physical function as part of this study. If you agree to wear a pedometer, you will wear the pedometer every day for a month during your waking hours. The pedometer used in the study is a small box that weighs less than an ounce and is smaller than a deck of playing cards. It is used to measure the number of steps you take during the day. Researchers will help you set the pedometer and show you how to use it. You will also keep a diary to record your use of the pedometer during this month. Researchers will meet with you during your clinic visits for chemotherapy at 2 weeks and 4 weeks to collect the data.

If you agree to take part in this study, you will have the following 4 types of study procedures performed:

Questionnaire:

Before chemotherapy that is scheduled by GI Medical Oncology Clinic starts, you will be asked to complete a questionnaire during a visit to the clinic. The questionnaire will measures physical and emotional symptoms. It should take about 5 minutes to finish. During this visit, the research staff will also teach you how to use the telephone system for measuring symptoms. You will tell the research staff the most convenient times for the telephone calls each week and the system will be set up to call you at that time.

Blood Draws:

Before you begin your chemotherapy treatments, you will have a sample of blood drawn (around 3½ tablespoons). The sample of blood will be used to measure levels of cytokines (biomarkers in the blood) and DNA (the genetic material in cells) in your blood before treatment starts. These cytokines may be related to symptoms experienced while having treatment for cancer.

You will have about 2½ tablespoons of blood drawn again when you complete first and second cycle of chemotherapy, and then at 2 months and 4 months after the start date of chemotherapy. Each blood sample will be drawn during your routine blood draw for continuing chemotherapy.

Symptoms Review:

You will have a MDASI-GI symptom assessment face to face, by regular mail, or through the phone calls. These will be used to measure symptom burden over time of the treatment and after treatment. The assessments will be done weekly for up to 4 months and then twice a month for up to an additional 14 months.

If your assessment is done by phone, it may be done by a study staff member or by using an interactive voice response telephone system (IVRS). During the study, the automated telephone system will call you once a week to ask you to rate your symptoms and how much the symptoms get in the way of your daily life. The information collected by these calls is only being used for this research study. This phone call should take about 5 minutes to complete.

This is an investigational study. Up to 100 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed cancer of the pancreas.
2. Patients must have inoperable locally advanced or metastatic disease.
3. Patients could be on treatment, or being planned for chemotherapy treatment.
4. Age 18 years of age or older
5. ECOG performance status 0-3
6. Ability to give consent in either English or Spanish

Exclusion Criteria:

1. Any condition (including unwillingness) that would impair the patient's ability to utilize the IVR system
2. Any recent surgical procedures (within 14 days, excluding biopsy, port-a-cath or picc line placement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will comprise 100 consecutive outpatients with metastatic disease being treated at the GI Medical Oncology clinic at M. D. Anderson.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-11-12 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Patient Reported Symptom Severity and Interference | Weekly for 8 cycles of chemotherapy, followed by twice a month for 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org